CLINICAL TRIAL: NCT01972230
Title: Sevoflurane Protective Effect on Ischemia Reperfusion Injury in Microvascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Ester Forastiere, director, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17713; Claudia (Registry Identifier: Claudia)
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Microvascular Breast Flap in Plastic Surgery
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bilanced group (Experimental): Sevofluorane adjusted to obtain an Et-Sevo of 1.8-2%, for all the time of the surgical procedure.
  Remifentanyl TCI adjusted according to protocol to maintain the range of 1-3 ng / ml.
  Interventions: Drug: Sevoflurane
- TCI group (Active Comparator): Propofol 3-4 mg / ml and remifentanyl 1-3 ng / ml according to protocol TCI
  Interventions: Drug: Diprivan + Remifentanil TCI

INTERVENTIONS:
Drug: Sevoflurane
  Arms: Bilanced group
Drug: Diprivan + Remifentanil TCI
  Arms: TCI group

SUMMARY:
This study aimed to evaluate the possible protective effect of anesthetic technique balanced (BAL) compared to total intravenous anesthetic technique (TIVA-TCI) in ischemia reperfusion injury in microvascular flap in plastic surgery. The investigators will evaluate the viability of the flap using tissue oximetry monitoring and the level of biochemical markers in a circle at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 yr
* ASA (American Society of Anesthesiology) I-II

Exclusion Criteria:

* Known unusual reaction to anesthetic drugs
* Evaluation of anesthesia increased risk for malignant hyperthermia.
* History of vascular disease.
* History of bleeding diathesis.
* Tabagism

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2013-01; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
tissutal oximetry average value of the flap measured with INVOS (In Vivo Optical Spectroscopy) system continuously. | 24 hours from the end of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Regina Elena Cancer Institute, Rome, RM, Italy